CLINICAL TRIAL: NCT03650088
Title: Adaptation of a Digital Weight Loss Intervention Promoting Self-regulation for Use in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-1078
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Results first posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus, Type 2; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Weight Loss Intervention (Experimental): Behavioral weight loss program with digital tools including smartphone app for dietary self-monitoring using a 'traffic light' approach, physical activity tracker, smart scale, and blood glucose monitoring plus with weekly consultation (in person or phone) with an interventionist for behavioral lessons and supports.
  Interventions: Behavioral: Behavioral weight loss with digital tools

INTERVENTIONS:
Behavioral: Behavioral weight loss with digital tools — Participants will monitor their diet in a study smart phone app using a 'traffic light' approach where foods are categorized as red (high fat and/or calorie), yellow (moderate fat/calorie, high nutrient), or green (low fat/calorie, high nutrient) and adhere to a red food limit recommendation, weigh daily on a digital scale whose data syncs to the study app, gradually increase physical activity and track it using a wearable device for which data is also synced to the app, and monitor blood glucose using Continuous Glucose Monitoring. Participants will meet weekly with a trained interventionist for behavioral lessons (adapted from Diabetes Prevention Program curriculum) and counseling.

SUMMARY:
The purpose of this study is to 1) adapt a weight loss app that the Tate team has previously developed to promote PA and diet and adapt them to the needs and perspectives of those with Type 2 Diabetes (T2DM), integrate daily monitoring of BG using continuous monitoring (CGM) and self-monitoring of diet using the simplified system, and develop appropriate displays of data to facilitate comprehension and decision making, 2) develop the modified intervention and, 3) conduct a pilot and feasibility study on short-term impacts of the intervention in overweight adult patients with T2DM not treated with medications in preparation for an R01 submission.

DETAILED DESCRIPTION:
Over 30 million Americans (nearly 10%) have diabetes, with the majority diagnosed with type 2 diabetes (T2D). The burden of T2D is costly with reduced quality of life, and increased morbidity, mortality, and health care expenditures. The majority of those with T2D are overweight, yet weight loss has been shown to be effective in the prevention and treatment of T2D.

In a 2017 Consensus Statement by the American Association of Clinical Endocrinologists and the American College of Endocrinology, the authors recommend weight loss of 5-10% for those with T2D whose BMI is > 25 kg/m^2 through comprehensive lifestyle intervention. Comprehensive lifestyle interventions are the gold standard in the behavioral treatment of obesity and diabetes. These evidence-based interventions include diet and physical activity prescriptions to reduce energy intake and increase expenditure; employ a variety of behavioral techniques to support these changes; and include in-person support from a multi-disciplinary team of interventionists. Changes in diet and activity as well as weight loss are essential for glycemic control in T2D. Lack of glycemic control leads to cardio- and micro-vascular complications that can significantly contribute to morbidity and mortality.

Self-regulation of behavior is an intervention approach to manage weight and to control blood glucose. Self-regulation involves having a goal, having access to information about whether the goal is being achieved, and if not, taking steps to restore equilibrium.

The intervention will be delivered through weekly in-person individual sessions and utilize a mobile phone app that integrates the diet, weight, physical activity and blood glucose data to support self-regulatory behaviors. In the first weekly session, participants will be oriented to the intervention and provided with their self-monitoring tools. They will be encouraged to weigh and track physical activity, Red foods and blood glucose (BG) daily and taught to use self-regulatory techniques for weight management and glycemic control. Similar to blood glucose self-regulation, participants are taught to compare the number on the scale each day to a standard or goal (weight loss goal) and, depending upon the comparison, make changes to their diet (i.e., Green foods or Red foods) or physical activity (i.e., moderate to vigorous physical activity (MVPA) or sedentary behavior(SB)) as needed. All participants will be given an initial weight loss goal of 5%.

Dietary Intervention

The specific recommendations for diet composition for T2D are consistent with the Traffic Light Diet concept and the investigators hypothesize that it can be used as a tool to encourage diet changes that will result in weight loss but will not be as burdensome as traditional calorie or carbohydrate monitoring methods. Rather than tracking calories as in traditional behavioral interventions, dietary goals and monitoring will be food-based. In the Traffic Light Diet, foods are categorized into Green, Yellow and Red categories. Users are encouraged to increase Green foods, moderate Yellow foods, and limit Red foods. Foods in the Green category include fruits, vegetables and certain very lean proteins, are low in calories, fat and sugar and rich in nutrients. The high volume, water content and fiber in fruits and vegetables and the protein from the lean meats and egg whites in this category help promote satiety while consuming fewer calories. The Yellow category includes moderately lean proteins, legumes, low fat dairy, whole grains, starchy vegetables, and low fat dressings. These foods are higher in calories than green food but are still a good source of nutrients. Red foods are high in calories, fat, and/or sugar and are not a good source of nutrients. The goal in the Traffic Light Diet is to increase Green foods and to limit Red foods. This emphasis on increasing healthful eating has been hypothesized to reduce feelings of deprivation and hunger. Participants in this study will be allowed unlimited Green foods.

Each participant will be given a personalized Red foods goal which will take into account baseline consumption of Red foods as well as baseline weight. During the formative evaluation, the investigators will be modifying the Red foods lists and goal recommendations based on patient and provider feedback. The underlying basis for the goal should result in a decrease in calories of 500-1000 per day which is consistent with standard behavioral treatment. Participants will only monitor Red foods to start. During individual counseling, interventionists will have the option to set a goal for Green foods and have the participant monitor those in the app if weight loss is not progressing as desired. Lesson content will model building healthy meals around green foods and participants will be provided with meal plans and recipes.

Physical Activity Intervention

The ultimate goal for the study will be to progress the participant to 150-200 minutes of moderate to vigorous physical activity. An initial goal will be based on baseline levels of PA as established during the first week of the study. Progression will occur each week based on individual progress of the participant. The participant will additionally focus on reductions in sedentary behavior with a study goal of exploring the feasibility of this alternative.

Study App

During the first individual session, the interventionist will work with the participant to download the app onto the participants' smartphone, familiarize them with the app, and set personal goals for weight, diet and physical activity, and BG monitoring.

Weight Goal and Monitoring--Participants will be provided a cell-enabled digital scale and instructed on setup and procedures for daily weighing.

Dietary Goal and Monitoring--Interventionists instruct on the Red foods list and monitoring of Red foods in the app. They will be instructed on portion size estimation and self-monitoring best practices (timing proximal to consumption). During the first week, participants will be advised to follow their normal diet in order to establish a baseline intake of Red foods. In the second session, the interventionist will work with the participant to set an initial Red foods goal.

Physical Activity Goal and Monitoring--Participants will be provided with a digital activity tracker and will set up the device and the app to allow for data transfer. Based on baseline physical activity from the first week of monitoring, the interventionist will work with the participant to set a goal for weekly physical activity minutes. Participants will also be advised on using the activity tracker to monitor sedentary time and to target sedentary behavior throughout the day.

BG Goals and Monitoring--Participants will be provided with an a Continuous Glucose Monitoring (CGM) unit. Recent advances in technology have made CGM much less invasive and simplified, thereby allowing for a better picture of glucose control given the number of data points available without the burden that previous CGM units presented. The interventionist will work with the participant to set goals for monitoring and ensure comprehension of CGM procedures.

Feedback: The app will provide text and graphic feedback comparing goals to behaviors and encourages adherence to the goals of daily weighing, monitoring and meeting Red foods and physical activity goals, and feedback on BG. For the purposes of this study, more rigorous intervention feedback will be delivered by the interventionist at weekly sessions.

Behavioral Lessons

A standard behavioral intervention based on the Diabetes Prevention Program (DPP) will be adapted for this protocol. Behavioral weight control approaches are founded on teaching skills and providing the support necessary to enable participants to adhere to the diet and physical activity prescription in their intervention. For the dietary intervention, materials will be adapted to reflect the Traffic Light Diet focus and modules for decreasing sedentary behavior will be added to those for increasing MVPA. Materials will be adapted with a focus on T2D. Lessons will be presented within the app and also available on paper at the individual counseling session. Brief review of the content will be done to assess comprehension and to explore personal applications.

Coaching Support

Individual counseling sessions will be semi-structured and led by Master's level or higher interventionists trained in behavioral weight control. Sessions typically last 30-45 minutes. Interventionists will review food, weight and activity progress through an administrative portal prior to individual sessions. During the weekly session, the interventionist will review self-monitoring records with the participant, set weekly goals, review behavioral lesson content introduced in the app, facilitate problem solving of any barriers the participant is having, and adapt treatment recommendations based on the needs of the participant. During the pilot phase, interventionists will record notes on the session to collect process data that will inform the continuing adaptation of the app and intervention protocols. This process data will also help to inform algorithms which will be developed in future studies to standardize counseling protocols for remote delivery and also to automate feedback in the app with the goal of broader dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 diabetes managed with lifestyle or pre-diabetes
* HBA1c >= 5.7%
* BMI 25 - 40 kg/m^2
* English speaking and writing
* not adhering the American College of Sports Medicine recommendation of 150 minutes of MVPA/week
* have a smartphone with internet access

Exclusion Criteria:

* current participation in another physical activity or weight control program
* report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q; items 1-4)
* substance abuse or mental health problems that would make it difficult to adhere to the dietary prescription
* moving out of the area during the study period
* unable to attend weekly sessions
* diagnosis of an eating disorder such as bulimia or anorexia
* currently pregnant, pregnant within the past 6 months, or planning to become pregnant within the next 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F. Tate, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through emails to individuals identified through medical records, informational emails, and social media posts and enrolled between October 2019 and October 2020 by research staff at the University of North Carolina at Chapel Hill Weight Research Program.
Period: Overall Study
Arm/Group | Weight Loss Intervention
Started | 18
Completed | 17
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Weight Loss Intervention
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (5.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Weight [Mean (Standard Deviation); unit: kg] | 94.97 (13.74)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.70 (4.20)
HbA1c Percent [Mean (Standard Deviation); unit: percent of total hemoglobin] | 6.45 (1.20)
Compliance Behavior and Efforts at Diabetes Self-Control [Mean (Standard Deviation); unit: units on a scale] — The Diabetes Locus of Control Scale assesses adherence to treatment recommendations for managing Type 2 diabetes; 18 items measured on a 6-point Likert scale where 1 is 'strongly disagree with the statement' and 6 is 'strongly agree with the statement'. Three subscales include internal locus of control (6 items), powerful others locus of control (6 items), and chance locus of control (6 items) and are calculated as the sum of values of the six responses for each subscale item with a range of 6-36 for each subscale. Higher values indicate higher attribution to the source of control.
  units on a scale
    Internal Locus of Control | 26.78 (3.08)
    Chance Locus of Control | 14.44 (4.07)
    Powerful Others Locus of Control | 17.67 (3.76)
Diabetes-related Quality of Life: The Diabetes Obstacles Questionnaire (DOQ-30) [Mean (Standard Deviation); unit: units on a scale] — The DOQ-30 assesses perceived hurdles to managing diabetes; 30 items each using a 5-point Likert-scale where 5 is strongly agree and 1 is strongly disagree. The scale includes nine subscales: 6 with 4 items (each ranging 4-20) and 3 with 2 items (each ranging 2-10). Subscale scores are calculated as the sum of individual subscale responses. Higher values indicate worse quality of life.
  units on a scale
    Relationships with Medical Professionals | 10.67 (2.59)
    Support from Family and Friends | 11.00 (3.41)
    Knowledge of the Disease | 10.94 (2.86)
    Lifestyle Changes | 8.50 (2.57)
    Exercising | 10.61 (2.77)
    Self-Monitoring | 10.28 (2.47)
    Uncertainty about a Consultation | 4.67 (1.03)
    Medication | 5.06 (1.95)
    Insulin-Use | 5.72 (1.74)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Weight will be measured on a digital scale
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Weight Loss Intervention
Number analyzed (Participants) | 17
kg | -4.54 (1.01)

2. Secondary Outcome: Change in Body Mass Index (BMI)
Description: BMI in kg/m^2
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Weight Loss Intervention
Number analyzed (Participants) | 17
kg/m^2 | -1.66 (0.39)

3. Secondary Outcome: Change in HbA1c Percent
Description: HbA1c will be measured by finger stick in the non-fasting state and analyzed using a point of care analyzer. HBA1c values 5.7 to 6.4% are considered pre-diabetes and 6.5% or higher are considered diabetes.
Time Frame: Baseline, Month 3
Population: At follow-up, 11 measurements were performed in clinic; 2 measurements were performed by the participant's Primary Care Provider and a report provided to the research staff; 4 participants had no data (due to COVID-19 restrictions, in person measurements were suspended)
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | Weight Loss Intervention
Number analyzed (Participants) | 13
percentage of total hemoglobin | -0.3 (0.08)

4. Secondary Outcome: Change in Compliance Behavior and Efforts at Diabetes Self-control
Description: The Diabetes Locus of Control Scale assesses adherence to treatment recommendations for managing Type 2 diabetes; 18 items measured on a 6-point Likert scale where 1 is 'strongly disagree with the statement' and 6 is 'strongly agree with the statement'. Three subscales include internal locus of control (6 items), powerful others locus of control (6 items), and chance locus of control (6 items) and are calculated as the sum of the six subscale item Likert-type responses with a range of 6-36 for each subscale. Higher values indicate higher attribution to the source of control.
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Weight Loss Intervention
Number analyzed (Participants) | 17
score on a scale
  Internal Locus of Control | -0.12 (1.01)
  Chance Locus of Control | -1.35 (0.67)
  Powerful Others Locus of Control | 0.65 (0.66)

5. Secondary Outcome: Change in Diabetes-related Quality of Life: The Diabetes Obstacles Questionnaire (DOQ-30)
Description: The Diabetes Obstacles Questionnaire (DOQ-30) assesses perceived obstacles to diabetes management: 30 items measured on a 5-point Likert-scale where 5 is strongly agree and 1 is strongly disagree. Nine subscales include relationships with medical professionals (4 items), support from friends and family (4 items), knowledge of the disease (4 items), lifestyle changes (4 items), exercising (4 items), self-monitoring (4 items), uncertainty about a consultation (2 items), medication (2 items), and insulin use (2 items). These are calculated as the sum of subscale responses with ranges of 4-20 for 4- item subscales and 2-10 for the 2- item subscales. Higher values indicate worse quality of life.
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Weight Loss Intervention
Number analyzed (Participants) | 17
score on a scale
  Relationships with Medical Professionals | -2.88 (0.70)
  Support from Friends and Family | -2.54 (0.61)
  Knowledge of the Disease | -4.06 (0.77)
  Lifestyle Changes | -1.24 (0.68)
  Exercising | -3.06 (0.66)
  Self-Monitoring | -2.29 (0.57)
  Uncertainty about a Consultation | -1 (0.30)
  Medication | -0.24 (0.47)
  Insulin use | -0.18 (0.42)

ADVERSE EVENTS:
Time Frame: From the time of informed consent through the Follow-Up assessment, a total of approximately 3 months.
Description: Adverse events were collected using the Medical Events Questionnaire at the follow-up assessment after the 12 week intervention.
Arm/Group | Weight Loss Intervention
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT03650088/Prot_SAP_ICF_000.pdf